CLINICAL TRIAL: NCT03610737
Title: A Multi-center, Randomized Controlled Study of the Vertos MILD Procedure With Conventional Medical Management Versus Conventional Medical Management Alone in the Treatment of Lumbar Spinal Stenosis.
Brief Title: The MOTION Study - Treatment of LSS With the MILD Procedure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vertos Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Motion
Record Dates: First submitted 2018-06-28; First posted 2018-08-01 (Actual); Results first posted 2023-05-01 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Spinal Stenosis, Lumbar Region, With Neurogenic Claudication
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MILD with CMM (Active Comparator): The MILD procedure is an image-guided minimally-invasive lumbar decompression with conventional medical managment
  Interventions: Device: MILD Procedure; Other: Conventional Medical Management (CMM)
- CMM alone (Active Comparator): Patient in the CMM alone group can have physical therapy, home exercise, pain medication, epidural steroid injections, nerve blocks, and other lumbar steroid injections.
  Interventions: Other: Conventional Medical Management (CMM)

INTERVENTIONS:
Device: MILD Procedure — The percutaneous procedure is performed under fluoroscopic guidance to effect a lumbar decompression with minimal surrounding tissue and bone disruption. The mild® Device Kit is utilized to access, capture and remove bone and tissue.
  Other Name: MILD lumbar decompression
  Arms: MILD with CMM
Other: Conventional Medical Management (CMM) — CMM can include physical therapy, home exercise, pain medication, epidural steroid injections, nerve blocks, and other lumbar steroid injections.

SUMMARY:
Prospective, multicenter, randomized controlled clinical study examining functional improvement in lumbar spinal stenosis (LSS) patients with neurogenic claudication who are treated with the MILD procedure plus conventional medical management (CMM) compared to those treated with CMM alone, as the control. Subjects in the control group are able to crossover and receive MILD after completion of 12-month follow-up. The study will provide objective functional improvement data for patients treated with the mild Procedure as first-line therapy in a real-world setting.

DETAILED DESCRIPTION:
The study will follow participants treated in the MILD plus CMM group and crossover participants for up to 5 years on annual bases.

ELIGIBILITY:
Inclusion Criteria:

* Patients experiencing neurogenic claudication symptoms for at least 3 months duration.
* LSS with neurogenic claudication
* Radiologic evidence of LSS with unilateral or bilateral ligamentum flavum ≥ 2.5mm confirmed by pre-op MRI or CT performed within 12 months of baseline visit.
* Patients with comorbid conditions commonly associated with spinal stenosis, such as osteophytes, facet hypertrophy, minor spondylolisthesis (Grade I without instability), foraminal stenosis, and/or disk protrusion may be included unless the treating physician has determined that the condition is too advanced.
* Stable opioid intake with no change during 30 days prior to enrollment.
* Available to complete all follow-up visits.

Exclusion Criteria:

* ODI Score < 31 (0-100 ODI Scale).
* NPRS Score < 5 (0-10 NPRS Scale).
* Lumbar epidural injections during eight weeks prior to study enrollment.
* Baseline analgesic medication greater than 90 milligram morphine equivalent (MME).
* Prior surgery at the same treatment level.
* Previously received interspinous spacer at the same treatment level.
* Previously received intradiscal procedure at the same treatment level.
* Previously received vertebral augmentation procedure at the same treatment level.
* Previously received the MILD procedure at the same treatment level.
* Received radiofrequency ablation at the same or the adjacent levels within 6 months prior to study enrollment.
* History of spinal fractures with current related pain symptoms.
* Grade II or higher spondylolisthesis.
* Motor deficit or disabling back and/or leg pain from causes other than LSS neurogenic claudication (e.g. acute compression fracture, metabolic neuropathy, or vascular claudication symptoms, etc.).
* Unable to walk ≥ 10 feet unaided before being limited by pain. In this context, 'unaided' means without the use of a cane, walker, railing, wall, another person or any other means of walking assistance.
* Previously randomized and/or treated in this clinical study.
* Epidural lipomatosis (if it is deemed to be a significant contributor of canal narrowing by the physician).
* On (or pending) Workman's Compensation or known to be considering litigation associated with back pain.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2025-04-30 (Estimated)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Newport Heache & Pain, Newport Beach, California
  - Centura Spine Center, Colorado Springs, Colorado
  - Spine & Pain Institute of Florida, Lakeland, Florida
  - SIMED, Ocala, Florida
  - The Pain Management and Rehabilitation Center, Seymour, Indiana
  - Kansas Pain Management, Overland Park, Kansas
  - Interventional Pain Management Specialists, Overland Park, Kansas
  - University of Kentucky, Lexington, Kentucky
  - MI Interventional Pain Center, Brownstown, Michigan
  - Michigan Pain Specialists, Ypsilanti, Michigan
  - Center for Pain Management, Hackensack, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Roanoke-Chowan Pain Management, Ahoskie, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - UH St. John Pain Management Center, Westlake, Ohio
  - Pennsylvania Pain & Spine Institute, Chalfont, Pennsylvania
  - Precision Spin Care, Tyler, Texas
  - The Center for Pain Relief, Charleston, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Deer TR, Chafin TB, Costandi SJ, Qu H, Kim C, Jassal N, Patel K, Calodney A. The MOTION study: Two-year results of a real-world randomized controlled trial of the mild(R) procedure for treatment of lumbar spinal stenosis. Pain Pract. 2024 Jan;24(1):109-119. doi: 10.1111/papr.13293. Epub 2023 Sep 3. PMID 37661347
- [Derived] Deer TR, Costandi SJ, Washabaugh E, Chafin TB, Wahezi SE, Jassal N, Sayed D. The MOTION Study: A Randomized Controlled Trial with Objective Real-World Outcomes for Lumbar Spinal Stenosis Patients Treated with the mild(R) Procedure: One-Year Results. Pain Med. 2022 Apr 8;23(4):625-634. doi: 10.1093/pm/pnac028. PMID 35167700

RESULTS

PARTICIPANT FLOW:
Groups:
- MILD With CMM: The MILD procedure is an image-guided minimally-invasive lumbar decompression with conventional medical managment
  MILD Procedure: The percutaneous procedure is performed under fluoroscopic guidance to effect a lumbar decompression with minimal surrounding tissue and bone disruption. The mild® Device Kit is utilized to access, capture and remove bone and tissue.
  Other Name: MILD lumbar decompression
  Conventional Medical Management (CMM): CMM can include physical therapy, home exercise, pain medication, epidural steroid injections, nerve blocks, and other lumbar steroid injections.
Period: Overall Study
Arm/Group | MILD With CMM | CMM Alone
Started | 77 | 78
Completed | 69 | 69
Not Completed | 8 | 9
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Death | 1 | 0
Not completed — Not treated | 5 | 2
Not completed — Missed Visit | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MILD With CMM | CMM Alone | Total
Number analyzed (Participants) | 77 | 78 | 155
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (7.4) | 66.8 (7.5) | 65.7 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 45 | 89
  Male | 33 | 33 | 66
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Oswestry Disability Index (ODI)
Description: Oswestry Disability Index (ODI) is a widely-used validated questionnaire use to measure a patient's functional disability. The total score ranges from 0 (no disability) - 100 (complete disability). Score categories: 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), 81-100 (bed bound or have an exaggerating).
Time Frame: Mean Change in Oswestry Disability Index (ODI) baseline to 12 month
Population: ODI Outcome Measure Mean Improvement
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MILD With CMM | CMM Alone
Number analyzed (Participants) | 69 | 69
score on a scale | 16.1 (19.0) | 2.0 (11.7)

ADVERSE EVENTS:
Time Frame: 1 Year
Description: Adverse events (AE) possibly related or definitely related to the study procedure will be collected for this study unless the AE is determined to be an SAE. All SAEs will be collected regardless of relationship, or lack thereof, to the study devices/procedures.
Arm/Group | MILD With CMM | CMM Alone
All-Cause Mortality (participants affected / at risk) | 1/77 | 0/78
Serious Adverse Events (participants affected / at risk) | 8/77 | 7/78
Other Adverse Events (participants affected / at risk) | 0/77 | 0/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MILD With CMM (N=77) | CMM Alone (N=78)
Cardiac disorders (Cardiac disorders) | 2 (3) | 0 (0)
General disorders (General disorders) | 1 (1) | 1 (1)
Infections and infestations (Infections and infestations) | 2 (2) | 2 (2)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2)
Nervous system disorders (Nervous system disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT03610737/Prot_SAP_000.pdf